CLINICAL TRIAL: NCT02310828
Title: The Efficacy of L-cysteine in Prevention of Cluster Headache. Randomized Intervention Trial With a Medical Device (Acetium® Capsules)
Brief Title: The Efficacy of L-cysteine in Prevention of Cluster Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biohit Oyj (Industry)
Collaborators: The Finnish Funding Agency for Technology and Innovation (TEKES) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-CLUSTPREV-1
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Cluster Headache
Keywords: Cluster headache; Migrainous neuralgia; Horton's headache; Histaminic cephalalgia
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetium (Experimental): Patient will administer Acetium capsules (100mg l-cysteine) twice a day for one month
  Interventions: Drug: Acetium
- Placebo (Placebo Comparator): Patient will administer placebo capsules twice a day for one month
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetium — Capsule for oral administration contains L-cysteine 100mg
  Other Names: Acetium capsule
  Arms: Acetium
Drug: Placebo — A placebo capsule matching Acetium for oral administration.
  Other Names: Acetium capsule placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to validate the novel hypothesis that daily use of L-cysteine (Acetium® capsules) is an effective means to decrease the frequency of (or completely abort) the attacks of cluster headache.

DETAILED DESCRIPTION:
Background: Cluster headache belongs to a group of idiopathic headache entities, the trigeminal autonomic cephalalgias (TACs), all of which involve short-lasting, unilateral, severe headache attacks and typical accompanying autonomic symptoms. The life-time prevalence of cluster headache for adults of all ages is around 125/100,000, or approximately 0.1%, with clear male dominance (4:1). Prophylactic treatment is an important part of the total management of cluster headache patients, having twofold goals: i) to reduce the frequency, painfulness, and/or duration of headache attacks, and ii) to increase the effectiveness of abortive therapy. During the past several decades, a large number of optional modalities have been tested as preventive measures of cluster headache. Not unexpectedly, the effects of any such preventive therapies are highly variable, and in many patients, the attack frequency is not under satisfactory control. Many of these drugs also have untoward side effects that offset their potential benefits.

Recently, spontaneous case testimonials were received by Biohit Oyj from migraine patients (and one with cluster headache) reporting that our new medical device, Acetium™ capsule (containing 100mg l-cysteine, developed for inactivation of acetaldehyde in the stomach contents after alcohol intake), proved to be highly effective against their headache attacks. Their attacks disappeared almost immediately after onset of L-cysteine administration, all of them remaining in complete remission for several months up to several years.

These spontaneous testimonials prompted us to formulate a novel study hypothesis that could possibly explain this dramatic effect of L-cysteine in prevention of headache attacks, to be tested in this RCT. This novel hypothesis is starting from the fact that, in cluster headache (a vascular-type of headache), swelling and dilatation of the blood vessels is necessary to provoke the attack.

It is known that Nitric Oxide (NO) is the final trigger of vascular headache attack, operating through phosphorylated protein kinase G (PKG) and Ca2+ channels, slowing the influx of calcium into the cell, which leads to smooth muscle relaxation and vasodilation. Histamine is a potent inducer of NO Synthase, making NO available locally on the vasculature, acting through endothelial H1-receptors. Histamine is synthesized from histidine in tissue mast cells, which are ubiquitous cells and their activation e.g. in the meninges has long been suspected to be involved in generating migraine headaches. Finally, one of the potent liberators of histamine from the mast cells is acetaldehyde, which, in turn, is effectively inactivated by L-cysteine (Acetium capsule). This led us to rational that by eliminating acetaldehyde in the stomach, L-cysteine could block (or reduce below the threshold levels) histamine liberation from the tissue mast cells and ECL cells in the stomach, thus arresting its multitude of functions, of which vasodilatation is critically involved in the cluster headache attack.

Objective: To validate the novel hypothesis that daily use of L-cysteine (Acetium capsules, 100mg twice a day) is an effective means to decrease the frequency of (or completely abort) the headache attacks in patients suffering from cluster headache.

Study design: A double-blind, randomized placebo-controlled multi-centre trial comparing Acetium capsules (100mg L-cysteine, twice a day) and placebo in prevention of headache attacks during a 1-month trial period. In brief, a cohort of 60 (up to100) voluntary subjects (women and men, with periodic or chronic cluster headache) are invited through the Finnish Migraine Association (FMA). To be eligible for the study, the subjects should: i) have the frequency of typical attacks up to 5 per day; ii) age between 18 and 65 years; and iii) have a minimum of co-morbidity. There are no restrictions on duration since the diagnosis, or the age at the onset of cluster headache. They should discontinue other prophylactic medication prior to study entry. Before enrolment, all subjects are requested to sign a written consent. The study protocol will be subjected for approval by the Committee on Medical Research Ethics (HUS).

Methods: The study setting is triple-blinded (participant-blind, investigator-blind, sponsor-blind). Placebo preparation with design and package identical to the test preparation will be used. Parallel group design instead of cross-over design is used. Randomization will be performed using a random number generator, with block size of 4, and stratified by gender.

The treatment period in both study arms will be 1 month. The participants should use (but accurately report) their usual symptomatic or acute treatment, because not anticipated to interfere with the study medication. During the 1-month treatment period, participants will be evaluated at weekly intervals by the study coordinator.

In addition to the baseline assessment of attack frequency, each subject will be requested to fill in a structured Questionnaire recoding their detailed headache history and other pertinent data on potential triggers. The headache diary is the main research tool used to monitor the efficacy of the test preparations, recording all predefined assessment measures (efficacy, tolerability and safety), and submitted to the study monitor on each FU visit.

In statistical analysis, both conventional techniques (e.g. non-parametric paired-samples and non-paired samples t-test), and more sophisticated methods will be used. The latter include i) life-table methods like Kaplan-Meier and Cox proportional hazards regression, as well as ii) generalized linear models (GEE and panel Poisson) and as a new technique in cluster headache RCTs, a competing risks regression to model the natural outcomes of the headache during the intervention. This study (n=60; the most modest scenario) is adequately powered (Type II error 0.80, type I error 0.05) to detect a true difference in attack frequency between 15 attacks/week in the placebo and 13.1 attacks/week in the Acetium arm. Given that the study subjects are enrolled among patients with typically 1-3 attacks/day, i.e., 7-21 (up to 35) attacks per week, and assuming a 10% reduction by placebo, there figures seem reasonable estimates for these power calculations.

Specific aims: The null hypothesis of the study implicates that l-cysteine is no better than placebo in prophylaxis of cluster headache during the 1-month intervention period. Rejection or not of the null hypothesis is based on comparison of the two arms for the primary study endpoint and (to lesser extent) for a series of secondary endpoints. The primary study endpoint (efficacy measure) is the number of attacks per week. Potentially useful secondary endpoints include: i) intensity of headache (4-tier nominal scale); ii) drug consumption for symptomatic or acute treatment; and iii) patients' preferences and satisfaction.

Study execution and time table: Meanwhile the final protocol is under evaluation for ethical approval by HUS, preparatory measures have been taken by informing the FMA about the planned study and asking their co-operation in encouraging the interested migraine patients to contact the study coordinator. Given the preliminary interest shown by the FMA, we are optimistic that the required cohort of volunteers can be enrolled within a short time, most likely by the end of 2013. However, because the subjects with episodic cluster headache must be enrolled during their on-going cluster episodes that typically follow a seasonal pattern, the enrolment of the total cohort (even n=60) inevitably needs to be completed over several months (up to one year).

Impact of the study: Given that L-cysteine is a natural (semi-essential) amino acid, converted to inert substance (MTCA) in the alimentary tract, it would comprise an ideal means to conduct prophylaxis of cluster headaches for years, without concern about the side effects that are inherent to many of the current treatment modalities. If the efficacy is proven in this formal RCT, the concept of using Acetium capsules in prophylactic treatment of cluster headache would represent a major step forward in a better clinical control of these frequently excruciating headaches.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years male/female
* episodic and chronic cluster headache
* the subjects should report cluster headache attacks with the frequency from one every second day up to five per day. The individual attacks should last from 15 minutes to 3h.

Exclusion Criteria:

* patients who meet the International Classification of Headache Disorders II criteria for medication overuse
* patients who have taken anti-psychotics or anti-depressant medications during the previous 3 months
* patients who abuse alcohol or other drugs
* potentially fertile and sexually active women who do not practise contraception
* other acute or chronic pain disorders
* severe psychiatric disease
* infections
* malignancy
* short life expectancy
* cardiovascular disease
* cerebrovascular disease
* uncontrolled hypertension
* degenerative central nervous system diseases
* pregnant and lactating women
* regular users of Acetium capsules for other indications
* renal dysfunction or cystinuria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-12-17 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
The frequency of headache attacks per week | 1 month
  The frequency of headache attacks per week, either during the entire treatment period or during the last treatment interval is compared with the baseline frequencies, to disclose differences between the two study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Mikko Kallela, MD, PhD, Principal Investigator — Helsinki Headache Center
Locations (6):
- Finland (6):
  - Terveystalo, Kamppi, Helsinki
  - Lääkärikeskus Aava, Helsingin Päänsärkykeskus Oy, Helsinki
  - Terveystalo, Jyväskylä, Jyväskylä
  - Terveystalo, Oulu, Oulu
  - Terveystalo, Tampere, Tampere
  - Terveystalo, Turku, Turku

IPD SHARING:
Plan to Share IPD: No